CLINICAL TRIAL: NCT00858143
Title: German Non Interventional Study For Patients Treated With Somavert®
Brief Title: Non Interventional Study For Patients Treated With Somavert®
Acronym: GPOS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A6291014
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Results first posted 2009-08-12 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-03

CONDITIONS: Acromegaly
Keywords: Open-label, national, prospective, observational, non-interventional, multi-center, post marketing surveillance study
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1
  Interventions: Other: Non Interventional Observation

INTERVENTIONS:
Other: Non Interventional Observation — Post marketing surveillance study = prospective, non-interventional observation of the use of Somavert®

SUMMARY:
This open-label, national, prospective, observational, non-interventional, multi-center, post marketing surveillance study was performed in order to examine the efficacy and safety of Somavert® in treatment of subjects with acromegaly and its effects on acromegaly related co-morbidities.

DETAILED DESCRIPTION:
Non probability samples

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosed acromegaly who were already being treated with Somavert® or were to start treatment with Somavert® were included in the study.

Exclusion Criteria:

* Subjects treated with an investigational drug for treatment of acromegaly.
* Subjects with symptoms such visual field loss, cranial nerve palsies or intracranial hypertension, indicating need for surgery.
* Women who were pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with diagnosed acromegaly who were already being treated with Somavert® or were to start treatment with Somavert® were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2004-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6291014&StudyName=Non%20Interventional%20Study%20For%20Patients%20Treated%20With%20Somavert%AE

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Somavert® (active ingredient: Pegvisomant 10/15/20 mg). Dose and schedule were at discretion of each treating physician. Safety evaluations based on all 311 patients who received at least one dose of Somavert® (safety set). Results from 270 patients in the intent-to-treat (ITT) population were analyzed to evaluate the efficacy of Somavert® therapy.
Groups:
- Somavert®: Somavert® 10/15/20 milligrams (mg)(active ingredient: Pegvisomant)
Period: Overall Study
Arm/Group | Somavert®
Started | 311 (Baseline)
Completed | 261
Not Completed | 50
Not completed — Adverse Event | 16
Not completed — Lack of Efficacy | 4
Not completed — Death | 7
Not completed — Other | 23

BASELINE CHARACTERISTICS:
Arm/Group | Somavert®
Number analyzed (Participants) | 311
Age Continuous [Mean (Standard Deviation); unit: years] | 50.3 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154
  Male | 157

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline Insulin-like Growth Factor I (IGF-I)
Description: Change: IGF-I concentration at observation minus IGF-I concentration at baseline (local laboratory, different assay).
Time Frame: Baseline, Follow-up 1 (FUP 1) at ~6 months , Follow-up 2 (FUP 2) at ~12 months, Follow-up 3 (FUP 3) at ~ 24 months, Follow-up 4 (FUP 4) at ~ 36 months, Follow-up 5 (FUP 5) at ~ 48 months, Follow-up 6 (FUP 6)at ~60 months
Population: Intent to Treat (ITT) Population, subjects who received at least one dose of Somavert during the observation period and had baseline and at least one post baseline efficacy measurement (n=number of subjects with efficacy measurement).
Measure: Mean (Standard Deviation); unit: micrograms per liter (ug/l)
Arm/Group | Somavert®
Number analyzed (Participants) | 270
micrograms per liter (ug/l)
  Follow-up 1 (n=243) | -200.3 (239.1)
  Follow-up 2 (n=202) | -202.6 (327.7)
  Follow-up 3 (n=131) | -273.7 (251.3)
  Follow-up 4 (n=71) | -319.6 (234.7)
  Follow-up 5 (n=18) | -296.6 (189.6)

2. Secondary Outcome: IGF-I Values Within Normal Range
Description: Number of participants who have IGF-I values within normal range (local laboratory, different assay).
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participant
Arm/Group | Somavert®
Number analyzed (Participants) | 270
participant
  Baseline (n=266) | 59
  Follow-up 1 (n=261) | 156
  Follow-up 2 (n=222) | 154
  Follow-up 3 (n=147) | 108
  Follow-up 4 (n=79) | 56
  Follow-up 5 (n=21) | 14

3. Secondary Outcome: IGF-I Values Above Normal Range
Description: Number of participants who have IGF-I values above normal range (local laboratory, different assay).
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participant
Arm/Group | Somavert®
Number analyzed (Participants) | 270
participant
  Baseline (n=266) | 207
  Follow-up 1 (n=261) | 105
  Follow-up 2 (n=222) | 68
  Follow-up 3 (n=147) | 39
  Follow-up 4 (n=79) | 23
  Follow-up 5 (n=21) | 7

4. Secondary Outcome: Change From Baseline Hemoglobin A 1c (HbA 1c)
Description: Change: HbA 1c at observation minus HbA 1c at baseline.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Somavert®
Number analyzed (Participants) | 270
percent (%)
  Follow-up 1 (n=124) | -0.3 (0.9)
  Follow-up 2 (n=123) | -0.3 (1.0)
  Follow-up 3 (n=80) | -0.3 (1.1)
  Follow-up 4 (n=41) | -0.3 (1.6)
  Follow-up 5 (n=10) | -0.0 (0.7)

5. Secondary Outcome: HbA 1c Values Within Normal Range
Description: Number of participants who have HbA 1c values within normal range.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participant
Arm/Group | Somavert®
Number analyzed (Participants) | 270
participant
  Baseline (n=173) | 104
  Follow-up 1 (n=132) | 85
  Follow-up 2 (n=127) | 78
  Follow-up 3 (n=82) | 57
  Follow-up 4 (n=43) | 30
  Follow-up 5 (n=10) | 7

6. Secondary Outcome: HbA 1c Values Below Normal Range
Description: Number of participants who have HbA 1c values below normal range.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5), 60 months (FUP 6)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Somavert®
Number analyzed (Participants) | 270
participants
  Baseline (n=173) | 0
  Follow-up 1 (n=132) | 1
  Follow-up 2 (n=127) | 1
  Follow-up 3 (n=82) | 1
  Follow-up 4 (n=43) | 0
  Follow-up 5 (n=10) | 0

7. Secondary Outcome: HbA 1c Values Above Normal Range
Description: Number of participants with HbA 1c values above normal range.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Somavert®
Number analyzed (Participants) | 270
participants
  Baseline (n=173) | 69
  Follow-up 1 (n=132) | 46
  Follow-up 2 (n=127) | 48
  Follow-up 3 (n=82) | 24
  Follow-up 4 (n=43) | 13
  Follow-up 5 (n=10) | 3

8. Secondary Outcome: Change From Baseline Glucose (Fasting)
Description: Change: glucose at observation minus glucose at baseline.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dl)
Arm/Group | Somavert®
Number analyzed (Participants) | 270
milligram per deciliter (mg/dl)
  Follow-up 1 (n=121) | -11.6 (39.6)
  Follow-up 2 (n=103) | -14.2 (40.1)
  Follow-up 3 (n=70) | -19.7 (45.7)
  Follow-up 4 (n=33) | -12.9 (51.0)
  Follow-up 5 (n=8) | -10.5 (18.3)

9. Secondary Outcome: Change From Baseline Glucose <(2 Hour Oral Glucose Tolerance Test (2h oGTT)>
Description: Change: glucose 2h oGTT at observation minus glucose 2h oGTT at baseline.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dl)
Arm/Group | Somavert®
Number analyzed (Participants) | 270
milligram per deciliter (mg/dl)
  Follow-up 1 (n=3) | -1.5 (38.7)
  Follow-up 2 (n=2) | -56.8 (85.4)
  Follow-up 3 (n=2) | -61.3 (79.0)

10. Secondary Outcome: Glucose Values Within Normal Range (Fasting)
Description: Number of participants who have glucose values within normal range (fasting).
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Somavert®
Number analyzed (Participants) | 270
participants
  Baseline (n=172) | 116
  Follow-up 1 (n=132) | 103
  Follow-up 2 (n=117) | 93
  Follow-up 3 (n=78) | 65
  Follow-up 4 (n=35) | 25
  Follow-up 5 (n=8) | 6

11. Secondary Outcome: Glucose Values Below Normal Range (Fasting)
Description: Number of participants with glucose values below normal range (fasting).
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Somavert®
Number analyzed (Participants) | 270
participants
  Baseline (n=172) | 2
  Follow-up 1 (n=132) | 3
  Follow-up 2 (n=117) | 1
  Follow-up 3 (n=78) | 1
  Follow-up 4 (n=35) | 0
  Follow-up 5 (n=8) | 0

12. Secondary Outcome: Glucose Values Above Normal Range (Fasting)
Description: Number of participants with glucose values above normal range (fasting).
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Somavert®
Number analyzed (Participants) | 270
participants
  Baseline (n=172) | 54
  Follow-up 1 (n=132) | 26
  Follow-up 2 (n=117) | 23
  Follow-up 3 (n=78) | 12
  Follow-up 4 (n=35) | 10
  Follow-up 5 (n=8) | 2

13. Secondary Outcome: Glucose (2 Hour Oral Glucose Tolerance Test (2h oGTT)) Values Within Normal Range
Description: Number of participants with glucose values (2h oGTT) within normal range.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Somavert®
Number analyzed (Participants) | 270
participants
  Baseline (n=7) | 5
  Follow-up 1 (n=4) | 3
  Follow-up 2 (n=3) | 3
  Follow-up 3 (n=3) | 3
  Follow-up 4 (n=0) | 0
  Follow-up 5 (n=0) | 0

14. Secondary Outcome: Glucose (2 Hour Oral Glucose Tolerance Test (2h oGTT)) Values Above Normal Range
Description: Number of participants with glucose values (2h oGTT) above normal range.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Somavert®
Number analyzed (Participants) | 270
participants
  Baseline (n=7) | 2
  Follow-up 1 (n=4) | 1
  Follow-up 2 (n=3) | 0
  Follow-up 3 (n=3) | 0
  Follow-up 4 (n=0) | 0
  Follow-up 5 (n=0) | 0

15. Secondary Outcome: IGF-I Absolute Values
Description: IGF-I absolute values (local laboratory, different assay).
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms per liter (ug/l)
Arm/Group | Somavert®
Number analyzed (Participants) | 270
micrograms per liter (ug/l)
  Baseline (n=252) | 480.1 (249.5)
  Follow-up 1 (n=243) | 277.2 (160.5)
  Follow-up 2 (n=202) | 281.6 (285.0)
  Follow-up 3 (n=131) | 240.6 (134.7)
  Follow-up 4 (n=71) | 236.1 (124.2)
  Follow-up 5 (n=18) | 241.8 (107.4)

16. Secondary Outcome: Absolute Glucose Values (Fasting)
Description: Absolute Glucose values (fasting)
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dl)
Arm/Group | Somavert®
Number analyzed (Participants) | 270
milligram per deciliter (mg/dl)
  Baseline (n=158) | 112.6 (44.3)
  Follow-up 1 (n=121) | 104.5 (42.6)
  Follow-up 2 (n=103) | 98.7 (34.0)
  Follow-up 3 (n=70) | 95.2 (17.6)
  Follow-up 4 (n=33) | 105.9 (42.7)
  Follow-up 5 (n=8) | 107.5 (31.1)

17. Secondary Outcome: Absolute Glucose Values (2h oGTT)
Description: Absolute Glucose values - 2 Hour Oral Glucose Tolerance Test (2h oGTT).
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dl)
Arm/Group | Somavert®
Number analyzed (Participants) | 270
milligram per deciliter (mg/dl)
  Baseline (n=5) | 130.6 (60.2)
  Follow-up 1 (n=3) | 145.3 (71.8)
  Follow-up 2 (n=2) | 108.1 (10.2)
  Follow-up 3 (n=2) | 112.6 (3.8)

18. Secondary Outcome: Absolute Hemoglobin A 1c (HbA 1c) Values
Description: Absolute value Hemoglobin A 1c (HbA 1c)
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Somavert®
Number analyzed (Participants) | 270
percent (%)
  Baseline (n=166) | 6.2 (1.2)
  Follow-up 1 (n=124) | 6.0 (1.1)
  Follow-up 2 (n=123) | 6.1 (1.1)
  Follow-up 3 (n=80) | 6.0 (1.1)
  Follow-up 4 (n=41) | 6.1 (1.1)
  Follow-up 5 (n=10) | 6.1 (0.9)

19. Secondary Outcome: Change From Baseline Insulin-Like Growth Factor I (IGF-I) in Diabetic Patients
Description: Change: IGF-I concentration at observation minus IGF-I concentration at baseline. (local laboratory, different assay).
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: micrograms per liter (ug/l)
Arm/Group | Somavert®
Number analyzed (Participants) | 192
micrograms per liter (ug/l)
  Follow-up 1 (n=75) | -207.5 [-263.6 to -151.3]
  Follow-up 2 (n=67) | -194.5 [-257.4 to -131.6]
  Follow-up 3 (n=44) | -274.6 [-353.9 to -195.4]
  Follow-up 4 (n=24) | -314.9 [-433.6 to -196.2]
  Follow-up 5 (n=4) | -90.5 [-348.8 to 167.74]

20. Secondary Outcome: Absolute Values Insulin-Like Growth Factor I (IGF-I) in Diabetic Patients
Description: Absolute values Insulin-Like Growth Factor I (IGF-I) in Patients with Diabetes (local laboratory, different assay).
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms per liter (ug/l)
Arm/Group | Somavert®
Number analyzed (Participants) | 192
micrograms per liter (ug/l)
  Baseline (n=78) | 478.8 (264.6)
  Follow-up 1 (n=75) | 276.4 (145.9)
  Follow-up 2 (n=67) | 293.2 (212.3)
  Follow-up 3 (n=44) | 239.3 (142.6)
  Follow-up 4 (n=24) | 242.5 (115.5)
  Follow-up 5 (n=4) | 311.3 (203.9)

21. Secondary Outcome: Insulin-Like Growth Factor I (IGF-I) Values Within Normal Range in Diabetic Patients
Description: Number of Diabetic Patients with Insulin-Like Growth Factor I (IGF-I) values Within Normal Range (local laboratory, different assay).
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Somavert®
Number analyzed (Participants) | 192
participants
  Baseline (n=81) | 14
  Follow-up 1 (n=80) | 41
  Follow-up 2 (n=74) | 47
  Follow-up 3 (n=49) | 35
  Follow-up 4 (n=26) | 16
  Follow-up 5 (n=5) | 3

22. Secondary Outcome: Insulin-Like Growth Factor I (IGF-I) Values Above Normal Range in Diabetic Patients
Description: Number of Diabetic Patients with Insulin-Like Growth Factor I (IGF-I) values Above Normal Range (local laboratory, different assay).
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Somavert®
Number analyzed (Participants) | 192
participants
  Baseline (n=81) | 67
  Follow-up 1 (n=80) | 39
  Follow-up 2 (n=74) | 27
  Follow-up 3 (n=49) | 14
  Follow-up 4 (n=26) | 10
  Follow-up 5 (n=5) | 2

23. Secondary Outcome: Absolute Values for Hemoglobin A 1c (HbA 1c) in Diabetic Patients
Description: Absolute Values for Hemoglobin A 1c (HbA 1c) in Patients with Diabetes
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Somavert®
Number analyzed (Participants) | 192
percent (%)
  Baseline (n=67) | 7.0 (1.4)
  Follow-up 1 (n=58) | 6.6 (1.2)
  Follow-up 2 (n=60) | 6.5 (1.2)
  Follow-up 3 (n=36) | 6.6 (1.3)
  Follow-up 4 (n=21) | 6.6 (1.3)
  Follow-up 5 (n=5) | 6.6 (1.0)

24. Secondary Outcome: Change From Baseline Hemoglobin A 1c (HbA 1c) in Diabetic Patients
Description: Change: HbA 1c at observation minus HbA 1c at baseline.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent (%)
Arm/Group | Somavert®
Number analyzed (Participants) | 192
percent (%)
  Follow-up 1 (n=58) | -0.4 [-0.8 to -0.1]
  Follow-up 2 (n=60) | -0.5 [-0.8 to -0.2]
  Follow-up 3 (n=36) | -0.5 [-1.0 to 0.0]
  Follow-up 4 (n=21) | -0.6 [-1.6 to 0.4]
  Follow-up 5 (n=5) | -0.2 [-1.3 to 0.9]

25. Secondary Outcome: HbA 1c Values Within Normal Range in Diabetic Patients
Description: Number of Diabetic Patients with HbA 1c Values Within Normal Range.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Somavert®
Number analyzed (Participants) | 192
participants
  Baseline (n=72) | 24
  Follow-up 1 (n=64) | 25
  Follow-up 2 (n=62) | 24
  Follow-up 3 (n=38) | 17
  Follow-up 4 (n=22) | 10
  Follow-up 5 (n=5) | 3

26. Secondary Outcome: HbA 1c Values Below Normal Range in Diabetic Patients
Description: Number of Diabetic Patients with HbA 1c Values Below Normal Range
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participant
Arm/Group | Somavert®
Number analyzed (Participants) | 192
participant
  Baseline (n=72) | 0
  Follow-up 1 (n=64) | 1
  Follow-up 2 (n=62) | 1
  Follow-up 3 (n=38) | 0
  Follow-up 4 (n=22) | 0
  Follow-up 5 (n=5) | 0

27. Secondary Outcome: HbA 1c Values Above Normal Range in Diabetic Patients
Description: Number of Diabetic Patients with HbA 1c Values Above Normal Range
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participant
Arm/Group | Somavert®
Number analyzed (Participants) | 192
participant
  Baseline (n=72) | 48
  Follow-up 1 (n=64) | 38
  Follow-up 2 (n=62) | 37
  Follow-up 3 (n=38) | 21
  Follow-up 4 (n=22) | 12
  Follow-up 5 (n=5) | 2

28. Secondary Outcome: Glucose Change From Baseline in Diabetic Patients (Fasting)
Description: Change: glucose at observation minus glucose at baseline
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milligram per deciliter (mg/dl)
Arm/Group | Somavert®
Number analyzed (Participants) | 192
milligram per deciliter (mg/dl)
  Follow-up 1 (n=42) | -17.2 [-35.6 to 1.1]
  Follow-up 2 (n=37) | -24.9 [-44.2 to -5.6]
  Follow-up 3 (n=21) | -50.7 [-81.4 to -20.0]
  Follow-up 4 (n=13) | -14.8 [-62.5 to 32.9]
  Follow-up 5 (n=3) | -17.7 [-76.7 to 41.3]

29. Secondary Outcome: Absolute Glucose Values in Diabetic Patients (Fasting)
Description: Absolute Glucose Values in Patients with Diabetes (fasting)
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dl)
Arm/Group | Somavert®
Number analyzed (Participants) | 192
milligram per deciliter (mg/dl)
  Baseline (n=51) | 142.1 (62.3)
  Follow-up 1 (n=42) | 131.0 (59.4)
  Follow-up 2 (n=37) | 112.9 (49.7)
  Follow-up 3 (n=21) | 101.9 (21.7)
  Follow-up 4 (n=13) | 130.6 (58.9)
  Follow-up 5 (n=3) | 120.7 (52.3)

30. Secondary Outcome: Glucose Values Within Normal Range in Diabetic Patients (Fasting)
Description: Number of Diabetic Patients (fasting) with Glucose Values Within Normal Range
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Somavert®
Number analyzed (Participants) | 192
participants
  Baseline (n= 57) | 24
  Follow-up 1 (n=47) | 28
  Follow-up 2 (n=42) | 25
  Follow-up 3 (n=25) | 18
  Follow-up 4 (n=14) | 6
  Follow-up 5 (n=3) | 2

31. Secondary Outcome: Glucose Values Above Normal Range in Diabetic Patients (Fasting)
Description: Number of Diabetic Patients (fasting) with Glucose Values Above Normal Range
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Somavert®
Number analyzed (Participants) | 192
participants
  Baseline (n=57) | 33
  Follow-up 1 (n=47) | 19
  Follow-up 2 (n=42) | 17
  Follow-up 3 (n=25) | 7
  Follow-up 4 (n=14) | 8
  Follow-up 5 (n=3) | 1

32. Secondary Outcome: Change in Headache Using Patient-assessed Acromegaly Symptom Questionnaire (PASQ)
Description: Change: score at observation minus score at baseline. Headache symptom in PASQ: disease-specific questionnaire consisting of 6 questions scoring 0-8. Maximum score indicates severe signs and symptoms, with lower scores reflecting improved quality of life.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4)
Population: ITT Population; subjects who received at least one dose of Somavert during the observation period and had baseline and at least one post baseline efficacy measurement (n=number of subjects with efficacy measurement). Data were available for 131 of the 270 ITT patients.
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Somavert®
Number analyzed (Participants) | 131
score on scale
  Follow-up 1 (n=107) | -0.3 [-0.7 to 0.1]
  Follow-up 2 (n=89) | -0.4 [-0.8 to 0.1]
  Follow-up 3 (n=60) | -0.2 [-0.6 to 0.2]
  Follow-up 4 (n=14) | -0.7 [-2.5 to 1.0]

33. Secondary Outcome: Change in Excessive Sweating Using Patient-assessed Acromegaly Symptom Questionnaire (PASQ)
Description: Change: score at observation minus score at baseline. Excessive sweating symptom in PASQ: disease-specific questionnaire consisting of 6 questions scoring 0-8. Maximum score indicates severe signs and symptoms, with lower scores reflecting improved quality of life.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4)
Population: as for outcome 32
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Somavert®
Number analyzed (Participants) | 131
score on scale
  Follow-up 1 (n=108) | -0.1 [-0.6 to 0.3]
  Follow-up 2 (n=89) | -0.4 [-0.9 to 0.2]
  Follow-up 3 (n=60) | -0.0 [-0.8 to 0.7]
  Follow-up 4 (n=14) | -0.8 [-2.8 to 1.3]

34. Secondary Outcome: Change in Joint Pain Using Patient-assessed Acromegaly Symptom Questionnaire (PASQ)
Description: Change: score at observation minus score at baseline. Joint pain symptom in PASQ: disease-specific questionnaire consisting of 6 questions scoring 0-8. Maximum score indicates severe signs and symptoms, with lower scores reflecting improved quality of life.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4)
Population: as for outcome 32
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Somavert®
Number analyzed (Participants) | 131
score on scale
  Follow-up 1 (n=108) | -0.6 [-1.0 to -0.2]
  Follow-up 2 (n=89) | -0.2 [-0.8 to 0.4]
  Follow-up 3 (n=60) | 0.0 [-0.5 to 0.6]
  Follow-up 4 (n=14) | 0.6 [-1.1 to 2.2]

35. Secondary Outcome: Change in Fatigue Using Patient-assessed Acromegaly Symptom Questionnaire (PASQ)
Description: Change: score at observation minus score at baseline. Fatigue symptom in PASQ: disease-specific questionnaire consisting of 6 questions scoring 0-8. Maximum score indicates severe signs and symptoms, with lower scores reflecting improved quality of life.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4)
Population: ITT Population; subjects who received at least one dose of Somavert during the observation period and had baseline and at least one post baseline efficacy measurement (n=number of subjects with efficacy measurement). Data were available for 130 of the 270 ITT patients.
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Somavert®
Number analyzed (Participants) | 131
score on scale
  Follow-up 1 (n=106) | 0.2 [-0.2 to 0.6]
  Follow-up 2 (n=88) | -0.5 [-0.9 to 0.0]
  Follow-up 3 (n=59) | -0.4 [-1.0 to 0.3]
  Follow-up 4 (n=14) | -0.4 [-1.6 to 0.8]

36. Secondary Outcome: Change in Soft Tissue Swelling Using Patient-assessed Acromegaly Symptom Questionnaire (PASQ)
Description: Change: score at observation minus score at baseline. Soft tissue swelling symptom in PASQ: disease-specific questionnaire consisting of 6 questions scoring 0-8. Maximum score indicates severe signs and symptoms, with lower scores reflecting improved quality of life.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4)
Population: as for outcome 32
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Somavert®
Number analyzed (Participants) | 131
score on scale
  Follow-up 1 (n=105) | -0.6 [-1.0 to -0.2]
  Follow-up 2 (n=88) | -0.8 [-1.4 to -0.2]
  Follow-up 3 (n=60) | -0.8 [-1.5 to -0.1]
  Follow-up 4 (n=14) | -1.2 [-3.1 to 0.6]

37. Secondary Outcome: Change in Numbness or Tingling of Limbs Using Patient-assessed Acromegaly Symptom Questionnaire (PASQ)
Description: Change: score at observation minus score at baseline. Numbness or tingling of limbs symptom in PASQ: disease-specific questionnaire consisting of 6 questions scoring 0-8. Maximum score indicates severe signs and symptoms, with lower scores reflecting improved quality of life.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4)
Population: as for outcome 35
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Somavert®
Number analyzed (Participants) | 131
score on scale
  Follow-up 1 (n=108) | -0.7 [-1.0 to -0.4]
  Follow-up 2 (n=89) | -0.6 [-1.0 to -0.2]
  Follow-up 3 (n=60) | -0.6 [-1.2 to -0.0]
  Follow-up 4 (n=14) | -0.8 [-2.0 to 0.4]

38. Secondary Outcome: Change in General Physical Condition Using Patient-assessed Acromegaly Symptom Questionnaire (PASQ)
Description: Change: score at observation minus score at baseline. General physical condition symptom in PASQ: disease-specific questionnaire based on the previous 6 questions which evaluated headache, excessive sweating, joint pain, fatigue, soft tissue swelling and numbness or tingling of limbs. Scoring 0-10 (0 = worst and 10 = best possible).
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4)
Population: as for outcome 32
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Somavert®
Number analyzed (Participants) | 131
score on scale
  Follow-up 1 (n=106) | -0.6 [-0.9 to -0.2]
  Follow-up 2 (n=89) | -0.6 [-1.1 to -0.2]
  Follow-up 3 (n=59) | -0.6 [-1.3 to 0.1]
  Follow-up 4 (n=14) | -0.5 [-2.2 to 1.2]

39. Secondary Outcome: Change in Total PASQ Score Using Patient-assessed Acromegaly Symptom Questionnaire (PASQ)
Description: Total PASQ score: total score calculated as sum of items 1-6; range is 0-48. Change from baseline calculated as total score at observation minus total score at baseline. PASQ: disease-specific questionnaire consisting of 6 questions scoring 0-8. Maximum score indicates severe signs and symptoms, with lower scores reflecting improved quality of life.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4)
Population: as for outcome 32
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Somavert®
Number analyzed (Participants) | 131
score on scale
  Follow-up 1 (n=107) | -2.3 [-3.7 to -0.9]
  Follow-up 2 (n=89) | -2.7 [-4.6 to -0.8]
  Follow-up 3 (n=60) | -2.0 [-4.4 to 0.5]
  Follow-up 4 (n=14) | -3.5 [-9.8 to 2.9]

40. Secondary Outcome: Mean Change From Baseline for Body Weight
Description: Change: body weight at observation minus body weight at baseline
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Somavert®
Number analyzed (Participants) | 270
kilogram (kg)
  Follow-up 1 (n=213) | 0.0 (5.2)
  Follow-up 2 (n=185) | 0.6 (6.0)
  Follow-up 3 (n=118) | 2.1 (7.4)
  Follow-up 4 (n=61) | 1.6 (7.7)
  Follow-up 5 (n=13) | 3.0 (8.4)

41. Secondary Outcome: Change From Baseline for Diastolic Blood Pressure (BP)
Description: Change: diastolic blood pressure at observation minus diastolic blood pressure at baseline
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters per mercury (mmHg)
Arm/Group | Somavert®
Number analyzed (Participants) | 270
millimeters per mercury (mmHg)
  Follow-up 1 (n=217) | -1.0 (11.0)
  Follow-up 2 (n=189) | -1.2 (13.0)
  Follow-up 3 (n=124) | -1.5 (13.4)
  Follow-up 4 (n=64) | 1.8 (15.2)
  Follow-up 5 (n=15) | 2.5 (15.1)

42. Secondary Outcome: Change From Baseline for Systolic Blood Pressure (BP)
Description: Change: systolic blood pressure at observation minus systolic blood pressure at baseline
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters Mercury (mmHg)
Arm/Group | Somavert®
Number analyzed (Participants) | 270
millimeters Mercury (mmHg)
  Follow-up 1 (n=217) | -0.1 (17.2)
  Follow-up 2 (n=189) | -2.9 (18.1)
  Follow-up 3 (n=124) | -4.3 (19.2)
  Follow-up 4 (n=65) | 2.1 (21.4)
  Follow-up 5 (n=15) | 8.4 (15.4)

43. Secondary Outcome: Change From Baseline in Ring Size
Description: Change from baseline: ring size at observation minus ring size at baseline
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Somavert®
Number analyzed (Participants) | 270
millimeters
  Follow-up 1 (n=99) | 0.2 (4.7)
  Follow-up 2 (n=82) | -0.8 (8.3)
  Follow-up 3 (n=37) | -0.3 (11.8)
  Follow-up 4 (n=16) | -6.1 (15.7)
  Follow-up 5 (n=2) | 0.0 (0.0)

44. Secondary Outcome: Adjusted Mean Dose of Somavert® Needed to Normalize the IGF-I Concentration in the Safety Population
Description: Adjusted Mean Dose of Somavert® needed to normalize IGF-I concentration during study while simultaneously adjusting for potential confounding baseline variables measured prior to Somavert® therapy. Multiple linear regression model used to evaluate dose needed to normalise IGF-I concentration. Model included terms for IGF-I, growth hormone, age, weight and gender.
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: The safety evaluations were based on all 311 patients who received at least one dose of Somavert® (safety set).
Measure: Number; unit: milligram (mg)
Arm/Group | Somavert®
Number analyzed (Participants) | 305
milligram (mg) | 16.8

45. Primary Outcome: Serious Adverse Events (SAE) and Adverse Events (AE)
Description: Long term safety of Somavert in treatment of patients with acromegaly
Time Frame: Baseline up to 5 years
Population: Safety Population; all patients who received at least one dose of Somavert® during the observation period.
Measure: Number; unit: participants
Arm/Group | Somavert®
Number analyzed (Participants) | 311
participants
  Serious Adverse Events (SAE's) | 116
  Adverse Events (AE's) | 197

46. Secondary Outcome: Adjusted Mean Dose of Somavert® Needed to Normalize the IGF-I Concentration in the ITT Population
Description: as for outcome 44
Time Frame: Baseline, 6 months (follow-up 1-FUP 1), 12 months (FUP 2), 24 months (FUP 3), 36 months (FUP 4), 48 months (FUP 5)
Population: Intent to Treat (ITT) Population, subjects who received at least one dose of Somavert during the observation period and had baseline and at least one post baseline efficacy measurement (n=number of subjects with efficacy measurement; n=129).
Measure: Number; unit: milligram (mg)
Arm/Group | Somavert®
Number analyzed (Participants) | 270
milligram (mg) | 16.4

ADVERSE EVENTS:
Arm/Group | Somavert®
Serious Adverse Events (participants affected / at risk) | 116
Other Adverse Events (participants affected / at risk) | 197
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Somavert®
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16/311
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7/311
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5/311
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/311
Pituitary tumour recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/311
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Extragonadal primary malignant teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Cholecystectomy (Surgical and medical procedures) | 8/311
Pituitary tumour removal (Surgical and medical procedures) | 8/311
Appendicectomy (Surgical and medical procedures) | 1/311
Cardiac pacemaker insertion (Surgical and medical procedures) | 1/311
Gallbladder operation (Surgical and medical procedures) | 1/311
Gastrectomy (Surgical and medical procedures) | 1/311
Hysterectomy (Surgical and medical procedures) | 1/311
Knee arthroplasty (Surgical and medical procedures) | 1/311
Knee operation (Surgical and medical procedures) | 1/311
Laparoscopic surgery (Surgical and medical procedures) | 1/311
Nephrectomy (Surgical and medical procedures) | 1/311
Pituitary gland radiotherapy (Surgical and medical procedures) | 1/311
Radiotherapy (Surgical and medical procedures) | 1/311
Radiotherapy to brain (Surgical and medical procedures) | 1/311
Umbilical hernia repair (Surgical and medical procedures) | 1/311
Hepatic enzyme increased (Investigations) | 13/311
Transaminases increased (Investigations) | 7/311
Insulin-like growth factor increased (Investigations) | 2/311
Alanine aminotransferase increased (Investigations) | 1/311
blood creatine phosphokinase increased (Investigations) | 1/311
Colonoscopy (Investigations) | 1/311
Gamma-glutamyltransferase increased (Investigations) | 1/311
Cholelithiasis (Hepatobiliary disorders) | 9/311
Bile duct stone (Hepatobiliary disorders) | 2/311
Biliary colic (Hepatobiliary disorders) | 2/311
Cholangitis (Hepatobiliary disorders) | 2/311
Hepatocellular injury (Hepatobiliary disorders) | 2/311
Cholecystitis (Hepatobiliary disorders) | 1/311
Cholecystitis acute (Hepatobiliary disorders) | 1/311
Pancreatitis (Gastrointestinal disorders) | 3/311
Colitis (Gastrointestinal disorders) | 1/311
Colonic polyp (Gastrointestinal disorders) | 1/311
Diverticular perforation (Gastrointestinal disorders) | 1/311
Gastritis haemorrhagic (Gastrointestinal disorders) | 1/311
Ileus (Gastrointestinal disorders) | 1/311
Pancreatitis acute (Gastrointestinal disorders) | 1/311
Umbilical hernia (Gastrointestinal disorders) | 1/311
Femur fracture (Injury, poisoning and procedural complications) | 2/311
Joint dislocation (Injury, poisoning and procedural complications) | 2/311
Lower limb fracture (Injury, poisoning and procedural complications) | 2/311
Road traffic accident (Injury, poisoning and procedural complications) | 2/311
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1/311
Fall (Injury, poisoning and procedural complications) | 1/311
Hand fracture (Injury, poisoning and procedural complications) | 1/311
Rib fracture (Injury, poisoning and procedural complications) | 1/311
Whiplash injury (Injury, poisoning and procedural complications) | 1/311
Epilepsy (Nervous system disorders) | 3/311
Anosmia (Nervous system disorders) | 1/311
Cerebrospinal fistula (Nervous system disorders) | 1/311
Cerebrospinal fluid rhinorrhoea (Nervous system disorders) | 1/311
Chiasma syndrome (Nervous system disorders) | 1/311
Hypoaesthesia (Nervous system disorders) | 1/311
Hyposmia (Nervous system disorders) | 1/311
Reversible ischaemic neurological deficit (Nervous system disorders) | 1/311
Transient ischaemic attack (Nervous system disorders) | 1/311
Aortic valve incompetence (Cardiac disorders) | 2/311
Tachyarrhythmia (Cardiac disorders) | 2/311
Acute myocardial infarction (Cardiac disorders) | 1/311
Angina pectoris (Cardiac disorders) | 1/311
Aortic valve sclerosis (Cardiac disorders) | 1/311
Atrial fibrillation (Cardiac disorders) | 1/311
Cardiac failure (Cardiac disorders) | 1/311
Coronary artery disease (Cardiac disorders) | 1/311
Cyanosis (Cardiac disorders) | 1/311
Myocardial infarction (Cardiac disorders) | 1/311
Ventricular fibrillation (Cardiac disorders) | 1/311
Ventricular tachycardia (Cardiac disorders) | 1/311
Cardiac death (General disorders) | 2/311
Application site necrosis (General disorders) | 1/311
Condition aggravated (General disorders) | 1/311
Disease progression (General disorders) | 1/311
No adverse event (General disorders) | 1/311
Pain (General disorders) | 1/311
Deep vein thrombosis (Vascular disorders) | 3/311
Hypertension (Vascular disorders) | 2/311
Hypertensive crisis (Vascular disorders) | 1/311
Peripheral circulatory failure (Vascular disorders) | 1/311
Adrenocortical insufficiency acute (Endocrine disorders) | 2/311
Toxic nodular goitre (Endocrine disorders) | 2/311
Hypopituitarism (Endocrine disorders) | 1/311
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2/311
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/311
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2/311
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1/311
Infection (Infections and infestations) | 2/311
Pneumonia (Infections and infestations) | 2/311
Back pain (Musculoskeletal and connective tissue disorders) | 1/311
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1/311
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1/311
Myalgia (Musculoskeletal and connective tissue disorders) | 1/311
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1/311
Diabetes mellitus (Metabolism and nutrition disorders) | 1/311
Diabetic foot (Metabolism and nutrition disorders) | 1/311
Electrolyte imbalance (Metabolism and nutrition disorders) | 1/311
Anaemia (Blood and lymphatic system disorders) | 1/311
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1/311
Blindness transient (Eye disorders) | 1/311
Optic ischaemic neuropathy (Eye disorders) | 1/311
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/311
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/311
Hydronephrosis (Renal and urinary disorders) | 1/311
Menorrhagia (Reproductive system and breast disorders) | 1/311
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Somavert®
Hepatic enzyme increased (Investigations) | 21/311
Transaminases increased (Investigations) | 11/311
Alanine aminotransferase increased (Investigations) | 4/311
Insulin-like growth factor increased (Investigations) | 3/311
Aspartate aminotransferase increased (Investigations) | 2/311
Gamma-glutamyltransferase increased (Investigations) | 2/311
Weight increased (Investigations) | 2/311
Analgesic drug level increased (Investigations) | 1/311
Blood creatine phosphokinase increased (Investigations) | 1/311
Blood pressure increased (Investigations) | 1/311
Colonoscopy (Investigations) | 1/311
Waist circumference increased (Investigations) | 1/311
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17/311
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7/311
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5/311
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/311
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/311
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/311
Pituitary tumour recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/311
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Extragonadal primary malignant teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/311
Cholecystectomy (Surgical and medical procedures) | 8/311
Pituitary tumour removal (Surgical and medical procedures) | 8/311
Radiotherapy (Surgical and medical procedures) | 5/311
Radiotherapy to brain (Surgical and medical procedures) | 2/311
Appendicectomy (Surgical and medical procedures) | 1/311
Cardiac pacemaker insertion (Surgical and medical procedures) | 1/311
Gallbladder operation (Surgical and medical procedures) | 1/311
Gastrectomy (Surgical and medical procedures) | 1/311
Hypophysectomy (Surgical and medical procedures) | 1/311
Hysterectomy (Surgical and medical procedures) | 1/311
Knee arthroplasty (Surgical and medical procedures) | 1/311
Knee operation (Surgical and medical procedures) | 1/311
Laparoscopic surgery (Surgical and medical procedures) | 1/311
Nephrectomy (Surgical and medical procedures) | 1/311
Pituitary gland radiotherapy (Surgical and medical procedures) | 1/311
Polypectomy (Surgical and medical procedures) | 1/311
Therapy regimen changed (Surgical and medical procedures) | 1/311
Umbilical hernia repair (Surgical and medical procedures) | 1/311
Fat tissue increased (General disorders) | 5/311
Injection site erythema (General disorders) | 5/311
Disease progression (General disorders) | 4/311
Cardiac death (General disorders) | 2/311
Fatigue (General disorders) | 2/311
Injection site hypertrophy (General disorders) | 2/311
Injection site reaction (General disorders) | 2/311
Injection site swelling (General disorders) | 2/311
Pain (General disorders) | 2/311
Adverse drug reaction (General disorders) | 1/311
Application site necrosis (General disorders) | 1/311
Condition aggravated (General disorders) | 1/311
Drug ineffective (General disorders) | 1/311
Facial pain (General disorders) | 1/311
Feeling cold (General disorders) | 1/311
Influenza like illness (General disorders) | 1/311
Injection site induration (General disorders) | 1/311
Injection site oedema (General disorders) | 1/311
Injection site pruritus (General disorders) | 1/311
No adverse event (General disorders) | 1/311
Ulcer (General disorders) | 1/311
Headache (Nervous system disorders) | 13/311
Epilepsy (Nervous system disorders) | 3/311
Hyposmia (Nervous system disorders) | 2/311
Sciatica (Nervous system disorders) | 2/311
Anosmia (Nervous system disorders) | 1/311
Carpal tunnel syndrome (Nervous system disorders) | 1/311
Cerebral infarction (Nervous system disorders) | 1/311
Cerebrospinal fistula (Nervous system disorders) | 1/311
Cerebrospinal fluid rhinorrhoea (Nervous system disorders) | 1/311
Chiasma syndrome (Nervous system disorders) | 1/311
Disturbance in attention (Nervous system disorders) | 1/311
Dysaesthesia (Nervous system disorders) | 1/311
Hypoaesthesia (Nervous system disorders) | 1/311
IIIrd nerve paralysis (Nervous system disorders) | 1/311
Memory impairment (Nervous system disorders) | 1/311
Polyneuropathy (Nervous system disorders) | 1/311
Reversible ischaemic neurological deficit (Nervous system disorders) | 1/311
Spinal cord compression (Nervous system disorders) | 1/311
Transient ischaemic attack (Nervous system disorders) | 1/311
Visual field defect (Nervous system disorders) | 1/311
Constipation (Gastrointestinal disorders) | 6/311
Pancreatitis (Gastrointestinal disorders) | 3/311
Diarrhoea (Gastrointestinal disorders) | 2/311
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2/311
Abdominal pain lower (Gastrointestinal disorders) | 1/311
Abdominal pain upper (Gastrointestinal disorders) | 1/311
Colitis (Gastrointestinal disorders) | 1/311
Colonic polyp (Gastrointestinal disorders) | 1/311
Diverticular perforation (Gastrointestinal disorders) | 1/311
Dyspepsia (Gastrointestinal disorders) | 1/311
Faecal incontinence (Gastrointestinal disorders) | 1/311
Gastric cyst (Gastrointestinal disorders) | 1/311
Gastritis (Gastrointestinal disorders) | 1/311
Gastritis erosive (Gastrointestinal disorders) | 1/311
Gastritis haemorrhagic (Gastrointestinal disorders) | 1/311
Gastrointestinal pain (Gastrointestinal disorders) | 1/311
Gingivitis (Gastrointestinal disorders) | 1/311
Haemorrhoids (Gastrointestinal disorders) | 1/311
Ileus (Gastrointestinal disorders) | 1/311
Nausea (Gastrointestinal disorders) | 1/311
Pancreatitis acute (Gastrointestinal disorders) | 1/311
Reflux oesophagitis (Gastrointestinal disorders) | 1/311
Stomach discomfort (Gastrointestinal disorders) | 1/311
Umbilical hernia (Gastrointestinal disorders) | 1/311
Cholelithiasis (Hepatobiliary disorders) | 13/311
Biliary colic (Hepatobiliary disorders) | 3/311
Bile duct stone (Hepatobiliary disorders) | 2/311
Cholangitis (Hepatobiliary disorders) | 2/311
Hepatocellular injury (Hepatobiliary disorders) | 2/311
Cholecystitis (Hepatobiliary disorders) | 1/311
Cholecystitis acute (Hepatobiliary disorders) | 1/311
Hepatic cyst (Hepatobiliary disorders) | 1/311
Adrenal insufficiency (Endocrine disorders) | 3/311
Hypopituitarism (Endocrine disorders) | 3/311
Adrenocortical insufficiency acute (Endocrine disorders) | 2/311
Gonadotrophin deficiency (Endocrine disorders) | 2/311
Hypogonadism (Endocrine disorders) | 2/311
Toxic nodular goitre (Endocrine disorders) | 2/311
Diabetes insipidus (Endocrine disorders) | 1/311
Hyperparathyroidism primary (Endocrine disorders) | 1/311
Hyperprolactinaemia (Endocrine disorders) | 1/311
Hyperthyroidism (Endocrine disorders) | 1/311
Pituitary haemorrhage (Endocrine disorders) | 1/311
Secondary hypothyroidism (Endocrine disorders) | 1/311
Hypertension (Vascular disorders) | 12/311
Deep vein thrombosis (Vascular disorders) | 3/311
Hypertensive crisis (Vascular disorders) | 1/311
Macroangiopathy (Vascular disorders) | 1/311
Peripheral circulatory failure (Vascular disorders) | 1/311
Thrombophlebitis superficial (Vascular disorders) | 1/311
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3/311
Back pain (Musculoskeletal and connective tissue disorders) | 2/311
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2/311
Myalgia (Musculoskeletal and connective tissue disorders) | 2/311
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/311
Bone pain (Musculoskeletal and connective tissue disorders) | 1/311
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1/311
Chondropathy (Musculoskeletal and connective tissue disorders) | 1/311
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/311
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/311
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1/311
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/311
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1/311
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1/311
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1/311
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1/311
Diabetes mellitus (Metabolism and nutrition disorders) | 3/311
Vitamin D deficiency (Metabolism and nutrition disorders) | 3/311
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2/311
Hyperlipidaemia (Metabolism and nutrition disorders) | 2/311
Iron deficiency (Metabolism and nutrition disorders) | 2/311
Diabetic foot (Metabolism and nutrition disorders) | 1/311
Electrolyte imbalance (Metabolism and nutrition disorders) | 1/311
Hyperuricaemia (Metabolism and nutrition disorders) | 1/311
Hypoglycaemia (Metabolism and nutrition disorders) | 1/311
Hypokalaemia (Metabolism and nutrition disorders) | 1/311
Lactose intolerance (Metabolism and nutrition disorders) | 1/311
Pneumonia (Infections and infestations) | 3/311
Infection (Metabolism and nutrition disorders) | 2/311
Sinusitis (Infections and infestations) | 2/311
Dermatophytosis (Infections and infestations) | 1/311
Helicobacter gastritis (Infections and infestations) | 1/311
Helicobacter infection (Infections and infestations) | 1/311
Herpes Zoster (Infections and infestations) | 1/311
Lobar pneumonia (Infections and infestations) | 1/311
Urinary tract infection (Infections and infestations) | 1/311
Viral infection (Infections and infestations) | 1/311
Aortic valve incompetence (Cardiac disorders) | 2/311
Atrial fibrillation (Cardiac disorders) | 2/311
Cardiac failure (Cardiac disorders) | 2/311
Tachyarrhythmia (Cardiac disorders) | 2/311
Acute myocardial infarction (Cardiac disorders) | 1/311
Angina pectoris (Cardiac disorders) | 1/311
Aortic valve sclerosis (Cardiac disorders) | 1/311
Arrhythmia (Cardiac disorders) | 1/311
Coronary artery disease (Cardiac disorders) | 1/311
Cyanosis (Cardiac disorders) | 1/311
Myocardial infarction (Cardiac disorders) | 1/311
Sinus arrhythmia (Cardiac disorders) | 1/311
Ventricular fibrillation (Cardiac disorders) | 1/311
Ventricular tachycardia (Cardiac disorders) | 1/311
Femur fracture (Injury, poisoning and procedural complications) | 2/311
Joint dislocation (Injury, poisoning and procedural complications) | 2/311
Lower limb fracture (Injury, poisoning and procedural complications) | 2/311
Road traffic accident (Injury, poisoning and procedural complications) | 2/311
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1/311
Fall (Injury, poisoning and procedural complications) | 1/311
Hand fracture (Injury, poisoning and procedural complications) | 1/311
Procedural headache (Injury, poisoning and procedural complications) | 1/311
Radiation associated pain (Injury, poisoning and procedural complications) | 1/311
Rib fracture (Injury, poisoning and procedural complications) | 1/311
Whiplash injury (Injury, poisoning and procedural complications) | 1/311
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 4/311
Alopecia (Skin and subcutaneous tissue disorders) | 2/311
Erythema (Skin and subcutaneous tissue disorders) | 1/311
Hyperhidrosis (Injury, poisoning and procedural complications) | 1/311
Rash (Skin and subcutaneous tissue disorders) | 1/311
Rash pruritic (Skin and subcutaneous tissue disorders) | 1/311
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2/311
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/311
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2/311
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/311
Bronchial irritation (Respiratory, thoracic and mediastinal disorders) | 1/311
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1/311
Loss of libido (Psychiatric disorders) | 2/311
Depressed mood (Psychiatric disorders) | 1/311
Depression (Psychiatric disorders) | 1/311
Middle insomnia (Psychiatric disorders) | 1/311
Restlessness (Psychiatric disorders) | 1/311
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3/311
Gynaecomastia (Reproductive system and breast disorders) | 1/311
Menorrhagia (Reproductive system and breast disorders) | 1/311
Prostatism (Reproductive system and breast disorders) | 1/311
Visual acuity reduced (Eye disorders) | 2/311
Blindness transient (Eye disorders) | 1/311
Cataract (Eye disorders) | 1/311
Glaucoma (Eye disorders) | 1/311
Optic ischaemic neuropathy (Eye disorders) | 1/311
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 3/311
Diabetic nephropathy (Renal and urinary disorders) | 1/311
Hydronephrosis (Renal and urinary disorders) | 1/311
Renal arteriosclerosis (Renal and urinary disorders) | 1/311
Renal atrophy (Renal and urinary disorders) | 1/311
Renal cyst (Renal and urinary disorders) | 1/311
Anaemia (Blood and lymphatic system disorders) | 2/311
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1/311
Hypoacusis (Ear and labyrinth disorders) | 1/311
House dust allergy (Immune system disorders) | 1/311
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/311
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/311

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.